CLINICAL TRIAL: NCT01110525
Title: A Phase I, Double-blind, Randomised, Placebo-controlled, Two-cycle Crossover, Drug-drug Interaction Study to Investigate the Effects of AZD1981 Tablets 400 mg Twice Daily on the PK and PD of Oral Contraceptives in Healthy Female Volunteers
Brief Title: A Drug-drug Interaction Study to Investigate the Effects of AZD1981 on the Metabolism and Pharmacodynamics of Oral Contraceptives
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: D9830C00015; 2010-018864-18 (EudraCT Number)
Record Dates: First submitted 2010-04-01; First posted 2010-04-26 (Estimated); Last update posted 2010-11-18 (Estimated); Status verified 2010-11

CONDITIONS: Oral Contraceptives
Keywords: Phase I; Drug-drug interaction; Oral contraceptives; AZD 1981
MeSH Terms: interventions — AZD1981

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): AZD1981 + Oral contraceptive
  Interventions: Drug: AZD1981; Drug: Neovletta 21/28
- 2 (Placebo Comparator): Placebo + Oral contraceptive
  Interventions: Drug: Neovletta 21/28; Drug: Placebo AZD1981

INTERVENTIONS:
Drug: AZD1981 — 4X100 mg per oral, twice daily for 28 days
  Arms: 1
Drug: Neovletta 21/28 — Once daily with (21) or without (28) pause for bleeding.
Drug: Placebo AZD1981 — 4X100 mg per oral, twice daily for 28 days
  Arms: 2

SUMMARY:
The primary purpose of this study is to determine whether the treatment with AZD1981 will affect the metabolism of hormones included in oral contraceptives.

ELIGIBILITY:
Inclusion Criteria:

* Females of childbearing potential
* Use of Neovletta or Neovletta 28 minimum 3 months prior to enrolment.
* Willing to use a highly effective method of birth control, ie, double barrier method contraception.

Exclusion Criteria:

* Pregnancy and/or lactation or delivery/abortion within 6 months prior to randomisation.
* Any clinically significant disease or disorder.
* Any clinically relevant abnormal findings in physical examination.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of of EE and LNG by analysis of the AUC and Css,max. | PK sampling will be performed regularly during the study period of two months.

SECONDARY OUTCOMES:
Effect on LH, FSH, SHBG, progesterone, and E2 during the menstrual cycle: Serum concentrations of LH, FSH, SHBG, progesterone and E2 | PD sampling will be done at the end of treatment period 1 and 2.
Safety and tolerability of the combination: Adverse events, safety laboratory variables, pulse, blood pressure, electrocardiogram and physical examinations | Safety will be monitored continously and safety assessments will be made on several occasions throughout the whole study.
Steady state PK of 1981 in combo with oral contraceptives AUCτ, Css,max, time to Cmax during a dosing interval (tmax ss);apparent plasma clearance (CLss/F) of AZD1981(tmax ss) of EE and LNG; Morning Ctrough values of EE and LNG will be measured. | PK-sampling of AZD1981 wil be done at the end of treatment period 1 and 2.

CONTACTS AND LOCATIONS:
Overall Officials: Eva S Pettersson, Study Director — AstraZeneca R&D; Wolfgang Kühn, Principal Investigator — Quintiles AB, Phase I Services; Aslak Rautio, Principal Investigator — Quintiles Hermelinen AB
Locations (2):
- Sweden (2):
  - Research Site, Luleå
  - Research Site, Uppsala